CLINICAL TRIAL: NCT01002768
Title: A Trial Investigating the Hypoglycaemic Response to NN1250 in Subjects With Type 1 Diabetes
Brief Title: Comparison of Hypoglycaemic Response Between NN1250 and Insulin Glargine in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3538; U1111-1111-8843 (Other: WHO); 2008-008356-16 (EudraCT Number)
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Day 1-4: Once daily subcutaneous (under the skin) injection similar to 80% of individual basal insulin requirement. Day 5: Three times the individual basal insulin requirement.
  Arms: IDeg
Drug: insulin glargine — Day 1-4: Once daily subcutaneous (under the skin) injection similar to 80% of individual basal insulin requirement. Day 5: Three times the individual basal insulin requirement.
  Arms: IGlar

SUMMARY:
This trial iss conducted in Europe. The aim of this clinical trial is to evaluate the hypoglycaemic response (the response to low blood sugar) to NN1250 (insulin degludec) in subjects with type 1 diabetes.

The trial is designed as a two-period, crossover trial where the trial participant is randomised to one of two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Use of insulin glargine within 3 months prior to first dosing of investigational product in this trial
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted hypoglycaemic symptoms score at nadir plasma glucose concentration | Within 0-46 hours after last trial product administration

SECONDARY OUTCOMES:
Baseline-adjusted hypoglycaemic symptoms score at each level of plasma glucose | Within 0-46 hours after last trial product administration
Time from start of hypoglycaemic induction until each level of plasma glucose is reached | Within 0-46 hours after last trial product administration
Time to increase from nadir plasma glucose to a plasma glucose concentration of 3.9 mmol/L | Within 0-46 hours after last trial product administration
Hypoglycaemic symptoms score during recovery from hypoglycaemia | Within 0-46 hours after last trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Koehler G, Heller S, Korsatko S, Roepstorff C, Rasmussen S, Haahr H, Pieber TR. Insulin degludec is not associated with a delayed or diminished response to hypoglycaemia compared with insulin glargine in type 1 diabetes: a double-blind randomised crossover study. Diabetologia. 2014 Jan;57(1):40-9. doi: 10.1007/s00125-013-3056-0. Epub 2013 Sep 22. PMID 24057153
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com